CLINICAL TRIAL: NCT01843790
Title: A Phase 2a, Placebo-Controlled, Randomized, Single-Blind Study of Weekly Doses of GCS-100 in Patients With Chronic Kidney Disease
Brief Title: A Phase 2a Study of Weekly Doses of GCS-100 in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCS-100-CS-4002
Record Dates: First submitted 2013-04-25; First posted 2013-05-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — GCS-100; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo, saline (Placebo Comparator): Saline, dosed weekly for 8 weeks
  Interventions: Drug: Placebo, Saline
- GCS-100 low dose (Experimental): Low dose of GCS-100 given IV once per week for 8 weeks
  Interventions: Drug: GCS-100
- GCS-100 high dose (Experimental): High dose of GCS-100 given IV once per week for 8 weeks
  Interventions: Drug: GCS-100

INTERVENTIONS:
Drug: GCS-100 — The amount (in mg) of GCS-100 to be administered will be determined based on body surface area, which will be calculated based on body weight and height. The study drug dose should be calculated on Day 1. Drug should be added to an infusion bag or syringe containing 0.9% Sodium Chloride Injection, USP. Drug be infused into a large vein via a large bore catheter to avoid local irritation and administered at no more than 2 mg/mL in no less than 60 mL.
  Arms: GCS-100 high dose; GCS-100 low dose
Drug: Placebo, Saline — The amount (in mg) of drug to be administered will be determined based on body surface area, which will be calculated based on body weight and height. The drug dose should be calculated on Day 1. Drug should be added to an infusion bag or syringe containing 0.9% Sodium Chloride Injection, USP. Drug be infused into a large vein via a large bore catheter to avoid local irritation and administered at no more than 2 mg/mL in no less than 60 mL.
  Other Names: Saline solution; 0.9% Sodium Chloride Injection
  Arms: Placebo, saline

SUMMARY:
The primary objective of this study is to compare the change in estimated glomerular filtration rate (eGFR) from baseline to Week 8 between placebo and GCS-100 treatment. The secondary objective is to determine the safety and tolerability of GCS-100 administered for 8 weeks relative to placebo. In addition, the study will measure the effect of GCS-100 on circulating galectin-3 and other markers of disease activity.

DETAILED DESCRIPTION:
Galectin-3 contributes to fibrosis, is elevated in patients with ESRD, and correlates with adverse outcomes (de Boer et. al., 2011, Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). Animal models with genetic knockout of galectin-3 demonstrate a reduction in structural and functional deficits in the kidney (Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). GCS-100 is a galectin- 3 antagonist that has been shown to reduce fibrosis pre-clinically. Based on the role of galectin-3 and fibrosis in kidney disease, the Sponsor believes GCS-100 may be effective at treating patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of understanding the purpose and risks of the study and is able to provide written informed consent
2. Subject is ≥18 and ≤75 years of age; patients >75 years old may be included at the request of the investigator and discretion of the Medical Monitor
3. Subject has an eGFR of 15 - 44 mL/min/1.73m2 determined using the 4-variable Modification of Diet in Renal Disease (MDRD) equation (see Section 10.1)
4. Patients with CKD diagnosis >12 months and stable, in the opinion of the investigator, within the past 3 months
5. Subject is willing and able to comply with all protocol requirements
6. Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least 1 year) and male subjects with partners of childbearing potential must agree to use medically acceptable methods of contraception throughout the study period

Exclusion Criteria:

1. Treatment with an experimental (unlicensed) drug within 4 weeks or ≤5 half-lives prior to screening
2. Kidney disease due to systemic lupus erythematosus (regardless of whether active or in remission), any form of vasculitis (regardless of whether active or in remission), IgA nephropathy, multiple myeloma, polycystic kidney disease, untreated obstructed nephropathy or any other causes that, in the opinion of the investigator, may put the subject at an increased risk
3. Planned renal replacement therapy of any kind within 6 months of randomization
4. Previous solid organ transplant
5. Systolic blood pressure ≤90 mmHg and ≥160 mmHg and diastolic blood pressure ≤40 mmHg and ≥100 mmHg at screening
6. Subject has clinical laboratory values of:

   1. Hemoglobin: ≤9 g/dL
   2. Total bilirubin: >1.5X the upper limit of normal (ULN)
   3. ALT and/or AST: >2.5X ULN
7. Current treatment with immunosuppressive agents, except for topical agents or inhaled steroids when conditions are chronic and stable
8. Treatment with any form of IV iron therapy within 4 weeks prior to screening
9. Known history of cancer (excluding non-melanoma skin cancer that is not being actively treated) within 5 years of screening
10. Known history of human immunodeficiency virus, active hepatitis C virus (HCV), active hepatitis B virus (HBV), or prior history of infection with HBV (HBcAb positive); if adequate hepatic function has been documented for patients with HCV or prior history of hepatitis B without evidence of cirrhosis, the Medical Monitor may approve their enrollment
11. Clinically relevant active infection and/or a serious co-morbid medical condition, such as recent myocardial infarction (within the last 6 months), unstable angina, difficult-to-control congestive heart failure, uncontrolled hypertension, difficult-to-control cardiac arrhythmias, severe or uncontrolled chronic obstructive or chronic restrictive pulmonary disease, and/or cirrhosis.
12. Subject had major surgery within 4 weeks of randomization
13. If female, subject is pregnant or breastfeeding
14. Subject has a concomitant disease or condition, including laboratory abnormalities, which, in the opinion of the investigator, could interfere with the conduct of the study or put the subject at unacceptable risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) from baseline relative to placebo after administration of GCS-100 for 8 weeks in patients with chronic kidney disease (CKD) and baseline eGFR of 15 - 44 mL/min/1.73m2 | 12 weeks

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability of GCS-100 administered for 8 weeks relative to placebo in patients with CKD | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Tidmarsh, MD, PhD, Study Director
Locations (4):
- United States (4):
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - California Institute of Renal Research, La Mesa, California
  - Denver Nephrology, Denver, Colorado
  - Clinical Advancement Center, PLLC, San Antonio, Texas